CLINICAL TRIAL: NCT06547125
Title: Multicenter, Evaluator-Blinded, Randomized, No-Treatment Controlled Study of the Effectiveness and Safety of JUVÉDERM® VOLITE™ Injectable Gel for the Improvement in Skin Quality
Brief Title: A Study to Assess Adverse Events and Effectiveness of Intradermally Injected JUVÉDERM® VOLITE™ Gel Filler in Adult Participants For the Improvement of Skin Quality
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M24-486
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Skin Quality Deficit
Keywords: Skin Quality Deficit; Juvederm Volite; AGN-8015

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JUVÉDERM® VOLITE™ (Experimental): Participants in the treatment group will receive a single dose at the study initiation. Participants are eligible for touch up treatment.
  Interventions: Device: JUVÉDERM® VOLITE™
- Control - No Treatment (Other): Participants in the control group will receive no treatment. At Month 2, these participants will have the option to receive the treatment.
  Interventions: Device: JUVÉDERM® VOLITE™; Other: Control

INTERVENTIONS:
Device: JUVÉDERM® VOLITE™ — Injection, intradermal
  Other Names: AGN-8015
Other: Control — No-treatment control
  Arms: Control - No Treatment

SUMMARY:
Facial fine lines and wrinkles are caused by skin thinning, loss of moisture, and loss of elasticity due to factors such as age, ultraviolet (UV) radiation, and environmental exposures. Today, many injectable fillers are used to treat facial aging and correct skin defects. In this study, adverse effects and effectiveness of JUVÉDERM® VOLITE™ will be assessed in the treatment of fine lines and improving skin quality.

VOLITE is an investigational device being developed for improving skin quality. In this study, participants are placed in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 3 chance that participants will be assigned to the no-treatment control group. Adult participants seeking improvement of skin quality, especially hydration and radiance, in the treatment area will be enrolled. Around 135 participants will be enrolled in the study at approximately 6 sites in China.

Participants in the treatment group will receive the initial injection of VOLITE; the control group will receive no treatment, but will have the opportunity to receive VOLITE after 2 months. Participants will be followed up for 12 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin types II-IV
* Participants' FACE-Q Satisfaction with Skin Scale scores must meet the following criteria:

  * Participants must have FACE-Q Satisfaction with Skin Scale sum of raw scores of 39 or less
  * Participants must score "Very Dissatisfied" or "Somewhat Dissatisfied" on the following two questions:

    * How hydrated your facial skin looks?
    * How radiant your facial skin looks?

Exclusion Criteria:

* Any skin condition in the face area that might not be suitable for injection
* Uncontrolled systemic disease
* History of anaphylactic shock, or allergy to lidocaine (or any amide-based anesthetics), hyaluronic acid (HA) products, or Streptococcal protein, or is planning to undergo desensitization therapy during the study
* Active autoimmune disease
* Tendency to develop hypertrophic scarring
* Currently undergoing chemotherapy/radiotherapy
* Is undergoing orthodontia before enrollment or is planning to undergo it during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status for Evaluating Investigator's (EI) Live Assessment of Global Aesthetic Improvement in Skin Quality on the Treatment Area Using the Global Aesthetic Improvement Scale (GAIS) | Month 2
  A "responder" is a participant who shows improvement in the overall aesthetic assessment on the treatment area using GAIS. GAIS is a 5-point scale ranging from 'Very Much Improved' to 'Worse'.
Number of Participants with Adverse Events (AEs) | Up to approximately Month 12
  An AE is defined as any untoward medical occurrence, unintended disease or injury, or any untoward clinical signs (including an abnormal laboratory finding) in participants, users, or other persons, whether or not related to the investigational medical device, and whether anticipated or unanticipated.

SECONDARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status for Participant's Assessment of Global Aesthetic Improvement in Skin Quality on the Treatment Area using GAIS | Month 2
  A "responder" is a participant who shows improvement in the overall aesthetic assessment in the treatment area using GAIS. GAIS is a 5-point scale ranging from 'Very Much Improved' to 'Worse'.
Percentage of Participants Achieving "Responder" Status for Treating Investigator's (TI) Assessment of Global Aesthetic Improvement of Skin Quality on the Treatment Area using GAIS | Month 2
  A "responder" is a participant who shows improvement in the overall aesthetic assessment in the treatment area using GAIS. GAIS is a 5-point scale ranging from 'Very Much Improved' to 'Worse'.
Change from Baseline on the Overall Score of FACE-Q Satisfaction with Skin Scale | Month 2
  The FACE Q Satisfaction with Skin is a validated 12-item scale that asks subjects to report their level of satisfaction with how their facial skin looked "in the past week." Response options are on a 4-point Likert scale ranging from Very dissatisfied to Very Satisfied. Total score is Rasch transformed from 0 (worst) to 100 (best).
Percentage of Participants with Responder Status based on EI's Live Assessments of Hydration Improvement on the Treatment Area Using the Aesthetic Improvement Scale for Hydration | Month 2
  A "responder" is a participant who shows aesthetic improvement in hydration of the treatment area ("Improved," "Much Improved," or "Very Much Improved" on the scale).
Percentage of Participants with Responder Status based on EI's Live Assessments of Radiance Improvement on the Treatment Area Using the Aesthetic Improvement Scale for Radiance | Month 2
  A "responder" is a participant who shows aesthetic improvement in radiance of the treatment area ("Improved," "Much Improved," or "Very Much Improved" on the scale).
Change from Baseline in Treatment Area Skin Elasticity Measurement | Month 2
  The trained designee will measure skin elasticity using the assigned instrument at the designated study visits.
Change from Baseline in Treatment Area Skin Hydration Measurement | Month 2
  The trained designee will measure skin hydration using the assigned instrument at the designated study visits.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (6):
- China (6):
  - China-Japan Friendship Hospital /ID# 260959, Beijing, Beijing Municipality
  - Peking University First Hospital /ID# 260957, Xicheng District, Beijing Municipality
  - Nanjing Drum Tower Hospital /ID# 260950, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University /ID# 260951, Nanjing, Jiangsu
  - Huashan Hospital, Fudan University /ID# 261582, Shanghai, Shanghai Municipality
  - Hangzhou First People's Hospital /ID# 260952, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-486